CLINICAL TRIAL: NCT00089895
Title: Early Glycoprotein IIb/IIIa Inhibition in Non-ST-segment Elevation Acute Coronary Syndrome: A Randomized, Placebo-Controlled Trial Evaluating the Clinical Benefits of Early Front-loaded Eptifibatide in the Treatment of Patients With Non-ST-segment Elevation Acute Coronary Syndrome (EARLY ACS)
Brief Title: EARLY ACS: Early Glycoprotein IIb/IIIa Inhibition in Patients With Non-ST-segment Elevation Acute Coronary Syndrome (Study P03684AM2)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03684
Record Dates: First submitted 2004-08-17; First posted 2004-08-19 (Estimated); Results first posted 2009-12-21 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Ischemia; Acute Coronary Syndrome
Keywords: myocardial infarction; acute coronary syndrome; non-ST-segment elevation; eptifibatide; Integrilin; glycoprotein IIb/IIIa inhibitor (GP IIb/IIIa); percutaneous coronary intervention (PCI); coronary artery bypass graph surgery (CABG); catheterization; angina; ischemia; cardiac ischemia; cardiovascular disease
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome; Myocardial Infarction; Angina Pectoris; Ischemia; Coronary Artery Disease; Cardiovascular Diseases | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eptifibatide (Experimental): Eptifibatide in addition to standard of care such as standard doses of aspirin, unfractionated heparin or low-molecular-weight heparin.
  Interventions: Drug: Eptifibatide (Integrilin)
- Placebo (Placebo Comparator): Placebo in addition to standard of care such as standard doses of aspirin, unfractionated heparin or low-molecular-weight heparin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eptifibatide (Integrilin) — intravenous; 180 mcg/kg bolus followed by infusion of 2 mcg/kg/min for 12 to 96 hours (or longer if necessary to complete the 18- to 24-hour post-PCI infusion period, or up to 120 hours in patients who proceed to CABG [coronary artery bypass graft]); second bolus of 180 mcg/kg administered 10 minutes after first bolus.
  Other Names: Integrilin; SCH 060936; SCH 60936
  Arms: Eptifibatide
Drug: Placebo — intravenous; delivery to match eptifibatide to maintain blind
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if early INTEGRILIN® (eptifibatide) therapy in patients with non-ST-segment elevation acute coronary syndrome (ACS) reduces the occurence of death, heart attack and urgent cardiac intervention (surgery) compared to placebo (with delayed provisional use of eptifibatide).

DETAILED DESCRIPTION:
This study will enroll patients who experience symptoms of acute coronary syndrome (experiencing chest pain at rest with episodes lasting at least 10 minutes) and who are planned to undergo invasive surgical procedures after being given study drug for 12 to 96 hours. There are two different treatment groups in this study; approximately half of the patients will go to each group and the likelihood of receiving study drug vs. placebo is 50/50 (like tossing a coin). Medications that are standard of care will be provided to the patients (all patients will be given aspirin and standard hospital doses of one of two other blood thinning drugs - unfractionated heparin (UFH) or low-molecular-weight heparin). Which one patients receive is at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent and comply with study procedures and follow-up through 1 year.
* Plan to undergo an invasive strategy after receiving study drug for 12 to 96 hours.
* Able to be randomized into the trial within 12 hours of having symptoms of acute coronary syndrome.
* Experiencing symptoms of cardiac ischemia at rest (angina or anginal equivalent) with episode(s) lasting at least 10 minutes and have at least 2 of the following:

  * 60 years of age or more
  * Electrocardiogram changes (ECG)
  * Elevated troponin (protein released in the blood stream in people suffering from acute coronary syndrome) or CK-MB levels
* Or have all 3 of the following:

  * Prior history of cardiovascular disease
  * Elevated troponin or CK-MB levels
  * 50-59 years of age

Exclusion Criteria:

* pregnancy (known or suspected)
* renal dialysis within 30 days prior to randomizing in study
* other serious illnesses or any condition that the investigator feels would pose a significant hazard to the patient if the investigational therapy was to be initiated
* Stroke (hemorrhagic stroke at any time or non-hemorrhagic stroke within previous 7 days), central nervous system damage (such as neoplasm, aneurysm, intracranial surgery), bleeding disorders (including gastrointestinal bleeding), or recent major surgery or major trauma.
* History of certain hematologic problems following treatment with heparin or eptifibatide.
* Therapy with certain related drugs within a short time before randomization into the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9406 (Actual)
Dates: Start 2004-11-01 (Actual); Primary Completion 2008-11-01 (Actual); Study Completion 2008-11-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Furtado RHM, Nicolau JC, Guo J, Im K, White JA, Sabatine MS, Newby LK, Giugliano RP. Morphine and Cardiovascular Outcomes Among Patients With Non-ST-Segment Elevation Acute Coronary Syndromes Undergoing Coronary Angiography. J Am Coll Cardiol. 2020 Jan 28;75(3):289-300. doi: 10.1016/j.jacc.2019.11.035. PMID 31976867
- [Derived] Farhan S, Clare RM, Jarai R, Giugliano RP, Lokhnygina Y, Harrington RA, Kristin Newby L, Huber K. Fasting glucose, NT-proBNP, treatment with eptifibatide, and outcomes in non-ST-segment elevation acute coronary syndromes: An analysis from EARLY ACS. Int J Cardiol. 2017 Apr 1;232:264-270. doi: 10.1016/j.ijcard.2017.01.007. Epub 2017 Jan 4. PMID 28089149
- [Derived] Kragholm K, Goldstein SA, Yang Q, Lopes RD, Schulte PJ, Bernacki GM, White HD, Mahaffey KW, Giugliano RP, Armstrong PW, Harrington RA, Tricoci P, Van de Werf F, Alexander JH, Alexander KP, Newby LK. Trends in Enrollment, Clinical Characteristics, Treatment, and Outcomes According to Age in Non-ST-Segment-Elevation Acute Coronary Syndromes Clinical Trials. Circulation. 2016 Apr 19;133(16):1560-73. doi: 10.1161/CIRCULATIONAHA.115.017299. Epub 2016 Mar 8. PMID 26957532
- [Derived] Kunadian V, Giugliano RP, Newby LK, Zorkun C, Guo J, Bagai A, Montalescot G, Braunwald E, Califf RM, Van de Werf F, Armstrong PW, Harrington R, Gibson CM. Angiographic outcomes with early eptifibatide therapy in non-ST-segment elevation acute coronary syndrome (from the EARLY ACS Trial). Am J Cardiol. 2014 Apr 15;113(8):1297-305. doi: 10.1016/j.amjcard.2014.01.404. Epub 2014 Jan 31. PMID 24607027
- [Derived] De Ferrari GM, Fox KA, White JA, Giugliano RP, Tricoci P, Reynolds HR, Hochman JS, Gibson CM, Theroux P, Harrington RA, Van de Werf F, White HD, Califf RM, Newby LK. Outcomes among non-ST-segment elevation acute coronary syndromes patients with no angiographically obstructive coronary artery disease: observations from 37,101 patients. Eur Heart J Acute Cardiovasc Care. 2014 Mar;3(1):37-45. doi: 10.1177/2048872613489315. Epub 2013 May 9. PMID 24562802
- [Derived] Kaul P, Tanguay JF, Newby LK, Hochman JS, Westerhout CM, Califf RM, Tricoci P, Gibson CM, Giugliano RP, Harrington RA, Van de Werf F, Armstrong PW. Association between bleeding and mortality among women and men with high-risk acute coronary syndromes: insights from the Early versus Delayed, Provisional Eptifibatide in Acute Coronary Syndromes (EARLY ACS) trial. Am Heart J. 2013 Oct;166(4):723-8. doi: 10.1016/j.ahj.2013.07.014. Epub 2013 Sep 5. PMID 24093853
- [Derived] Bagai A, White JA, Lokhnygina Y, Giugliano RP, Van de Werf F, Montalescot G, Armstrong PW, Tricoci P, Gibson CM, Califf RM, Harrington RA, Newby LK. Routine early eptifibatide versus delayed provisional use at percutaneous coronary intervention in high-risk non-ST-segment elevation acute coronary syndromes patients: an analysis from the Early Glycoprotein IIb/IIIa Inhibition in Non-ST-Segment Elevation Acute Coronary Syndrome trial. Am Heart J. 2013 Sep;166(3):466-73. doi: 10.1016/j.ahj.2013.05.019. Epub 2013 Jul 25. PMID 24016495
- [Derived] Klutstein MW, Westerhout CM, Armstrong PW, Giugliano RP, Lewis BS, Gibson CM, Lutchmedial S, Widimsky P, Steg PG, Dalby A, Zeymer U, Van de Werf F, Harrington RA, Newby LK, Rao SV. Radial versus femoral access, bleeding and ischemic events in patients with non-ST-segment elevation acute coronary syndrome managed with an invasive strategy. Am Heart J. 2013 Apr;165(4):583-590.e1. doi: 10.1016/j.ahj.2013.01.009. Epub 2013 Feb 22. PMID 23537976
- [Derived] Ezekowitz JA, Bakal JA, Westerhout CM, Giugliano RP, White H, Keltai M, Prabhakaran D, Tricoci P, Van de Werf F, Califf RM, Newby LK, Armstrong PW. The relationship between meteorological conditions and index acute coronary events in a global clinical trial. Int J Cardiol. 2013 Oct 3;168(3):2315-21. doi: 10.1016/j.ijcard.2013.01.061. Epub 2013 Feb 14. PMID 23416014
- [Derived] Pride YB, Mohanavelu S, Zorkun C, Kunadian V, Giugliano RP, Newby LK, Braunwald E, Califf RM, Harrington RA, Gibson CM; EARLY ACS Investigators. Association between angiographic complications and clinical outcomes among patients with acute coronary syndrome undergoing percutaneous coronary intervention: an EARLY ACS (Early Glycoprotein IIb/IIIa Inhibition in Non-ST-Segment Elevation Acute Coronary Syndrome) angiographic substudy. JACC Cardiovasc Interv. 2012 Sep;5(9):927-35. doi: 10.1016/j.jcin.2012.05.007. PMID 22995880
- [Derived] Piccini JP, White JA, Mehta RH, Lokhnygina Y, Al-Khatib SM, Tricoci P, Pollack CV Jr, Montalescot G, Van de Werf F, Gibson CM, Giugliano RP, Califf RM, Harrington RA, Newby LK. Sustained ventricular tachycardia and ventricular fibrillation complicating non-ST-segment-elevation acute coronary syndromes. Circulation. 2012 Jul 3;126(1):41-9. doi: 10.1161/CIRCULATIONAHA.111.071860. Epub 2012 May 29. PMID 22645292
- [Derived] Roe MT, White JA, Kaul P, Tricoci P, Lokhnygina Y, Miller CD, van't Hof AW, Montalescot G, James SK, Saucedo J, Ohman EM, Pollack CV Jr, Hochman JS, Armstrong PW, Giugliano RP, Harrington RA, Van de Werf F, Califf RM, Newby LK. Regional patterns of use of a medical management strategy for patients with non-ST-segment elevation acute coronary syndromes: insights from the EARLY ACS Trial. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):205-13. doi: 10.1161/CIRCOUTCOMES.111.962332. Epub 2012 Feb 28. PMID 22373905
- [Derived] Wang TY, White JA, Tricoci P, Giugliano RP, Zeymer U, Harrington RA, Montalescot G, James SK, Van de Werf F, Armstrong PW, Braunwald E, Califf RM, Newby LK. Upstream clopidogrel use and the efficacy and safety of early eptifibatide treatment in patients with acute coronary syndrome: an analysis from the Early Glycoprotein IIb/IIIa Inhibition in Patients with Non-ST-Segment Elevation Acute Coronary Syndrome (EARLY ACS) trial. Circulation. 2011 Feb 22;123(7):722-30. doi: 10.1161/CIRCULATIONAHA.110.958041. Epub 2011 Feb 7. PMID 21300952
- [Derived] Giugliano RP, White JA, Bode C, Armstrong PW, Montalescot G, Lewis BS, van 't Hof A, Berdan LG, Lee KL, Strony JT, Hildemann S, Veltri E, Van de Werf F, Braunwald E, Harrington RA, Califf RM, Newby LK; EARLY ACS Investigators. Early versus delayed, provisional eptifibatide in acute coronary syndromes. N Engl J Med. 2009 May 21;360(21):2176-90. doi: 10.1056/NEJMoa0901316. Epub 2009 Mar 30. PMID 19332455

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients in both treatment groups who were undergoing PCI could receive unblinded eptifibatide provisionally immediately before or during percutaneous coronary intervention (PCI) at the discretion of the investigator.
Groups:
- Eptifibatide: Eptifibatide in addition to standard of care which includes usage of aspirin, unfractionated heparin or low-molecular weight heparin.
- Placebo: Placebo in addition to standard of care which includes usage of aspirin, unfractionated heparin or low-molecular weight heparin.
Period: Overall Study
Arm/Group | Eptifibatide | Placebo
Started | 4722 (Number of Subjects Randomized with Intent to Treat) | 4684 (Number of Subjects Randomized with Intent to Treat)
Completed | 4687 (Number of Subjects treated) | 4642 (Number of Subjects treated)
Not Completed | 35 | 42
Not completed — Consent Withdrawn | 11 | 14
Not completed — Technical reason | 7 | 2
Not completed — Surgery | 0 | 1
Not completed — Bleeding | 0 | 2
Not completed — Physician Decision | 3 | 7
Not completed — Exclusion criteria met | 6 | 6
Not completed — Not otherwise specified | 4 | 8
Not completed — Missing | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eptifibatide | Placebo | Total
Number analyzed (Participants) | 4722 | 4684 | 9406
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10.6) | 66.7 (10.7) | 66.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1513 | 1462 | 2975
  Male | 3209 | 3222 | 6431

OUTCOME MEASURES:

1. Primary Outcome: Incidence of the Composite of Death, Myocardial Infarction (MI), Recurrent Ischemia Requiring Urgent Revascularization (RI-UR), and Thrombotic Bail-out.
Time Frame: 96 hours after randomization
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Eptifibatide | Placebo
Number analyzed (Participants) | 4722 | 4684
percentage of participants | 9.3 | 10.0

2. Secondary Outcome: Incidence of the Composite of Death/MI.
Time Frame: 30 days after randomization
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Eptifibatide | Placebo
Number analyzed (Participants) | 4722 | 4684
percentage of participants | 11.2 | 12.3

ADVERSE EVENTS:
Time Frame: Through hospital discharge or 120 hours after randomization, whichever occurred first.
Arm/Group | Eptifibatide | Placebo
Serious Adverse Events (participants affected / at risk) | 66/4686 | 60/4643
Other Adverse Events (participants affected / at risk) | 0/4686 | 0/4643
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=4686) | Placebo (N=4643)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1)
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ADRENOCORTICAL INSUFFICIENCY ACUTE (Endocrine disorders) | 1 (1) | 0 (0)
OPHTHALMOPLEGIA (Eye disorders) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
IMPLANT SITE EFFUSION (General disorders) | 1 (1) | 0 (0)
INJECTION SITE PAIN (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 2 (2)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
HEPATITIS A (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PERIRECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 5 (5) | 8 (8)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 3 (3)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRAIN OEDEMA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1)
PARKINSONISM (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 2 (2)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 1 (1)
IGA NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHRITIS INTERSTITIAL (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROSCLEROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 6 (6) | 4 (4)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 6 (6) | 5 (5)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 (2) | 0 (0)
RENAL INFARCT (Renal and urinary disorders) | 0 (0) | 1 (1)
ANOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PLEURAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
AORTIC DISSECTION (Vascular disorders) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less